CLINICAL TRIAL: NCT03160040
Title: Retrospective, Observational Evaluation of the Utilization, Outcomes, and Adverse Events Associated With Minocin IV for the Treatment of Infections Presumed or Confirmed to be Caused by Gram-negative Bacteria in a Real World Setting
Brief Title: A Retrospective Observational Study to Evaluate the Utilization, Outcomes, and Adverse Events in Participants Treated With Minocin® (Minocycline) for Infections Caused by Gram-negative Bacteria in a Real World Setting
Status: Completed | Type: Observational
Sponsor: Rempex (a wholly owned subsidiary of Melinta Therapeutics, Inc.) (Industry)
Responsible Party: Sponsor
Organization: Melinta Therapeutics, Inc. (Industry)
Other Study IDs: MDCO-MIN-16-05
Record Dates: First submitted 2017-05-17; First posted 2017-05-19 (Actual); Last update posted 2023-08-28 (Actual); Status verified 2023-08

CONDITIONS: Gram-Negative Bacterial Infections
MeSH Terms: conditions — Gram-Negative Bacterial Infections | interventions — Minocycline

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Minocycline IV: Participants who received 2 doses over 48 hours if given once daily or 4 doses over 48 hours if given twice daily of minocycline intravenous (IV) as monotherapy, with or without transition to oral minocycline.
  Interventions: Drug: Minocycline IV

INTERVENTIONS:
Drug: Minocycline IV — This study is an observational study. All participants were administered minocycline IV prior to enrollment in this study.
  Other Names: Minocin®

SUMMARY:
This study is a retrospective, observational study to evaluate minocycline use in participants under real world conditions.

DETAILED DESCRIPTION:
This study is a retrospective, observational study to evaluate minocycline use in participants under real world conditions.

ELIGIBILITY:
Inclusion Criteria:

* The participant was treated with Minocin IV for a presumed or culture-confirmed gram-negative infection, as monotherapy or part of a broader regimen, for at least 48 hours.
* The participant treatment for gram-negative infection was initiated May 1, 2015, or later.
* The participant was at least 18 years old.
* This was the first course of Minocin IV administered to the participant within the study period for the treatment of gram-negative infection.
* At least 60 days has elapsed since the participant received the last dose of Minocin IV therapy for a presumed or confirmed gram-negative infection (prior to data entry into the electronic case report form, including step-down to oral therapy.

Exclusion Criteria:

* The participant received Minocin IV as a part of a controlled clinical trial.
* The participant received Minocin IV as a part of a Medicines Company- or Rempex Company-sponsored pharmacoeconomic outcomes study.
* Pregnancy (in the participant's or participant's partner) occurred after the first dose of Minocin IV through hospital discharge.
* Female participants were pregnant or nursing at the time of enrollment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Participants in intensive care unit (ICU) and non-ICU real world settings throughout the United States, who received at least 48 hours of minocycline IV in the treatment of documented gram-negative infections.
Sampling Method: Probability Sample
Enrollment: 71 (Actual)
Dates: Start 2017-10-11 (Actual); Primary Completion 2018-05-01 (Actual); Study Completion 2018-05-01 (Actual)

PRIMARY OUTCOMES:
Number Of Participants With Each Gram-negative Bacterial Infection Being Treated With Minocycline IV | Day 1
  The types of primary infections refers to only presumed or documented gram-negative bacterial infections.
Infection-related Length Of Stay For Infections Being Treated With Minocycline IV | Up to 30 days after minocycline IV infusion
  Data will be collected to include infection-related length of stay , which is defined as the difference between the day of initiation of antimicrobial administration for the primary infection and day of discontinuation, death, or discharge date, whichever is sooner. This may include minocycline IV or other empiric antimicrobial regimen.
Number Of Participants With A Microbiologic Response | Up to 30 days after minocycline IV infusion
  The number of participants with a gram-negative pathogen for which minocycline IV is used for treatment of the primary infection site(s) and the number of participants with a gram-positive pathogen recovered from a secondary infection site or from a mixed culture also containing the targeted gram-negative pathogen will be presented.
Duration Of Treatment With Minocycline IV | Day 1 through end of infusion with minocycline
  The number of days of treatment with minocycline IV will be presented.
Use Of Concomitant Antibiotics With Minocycline IV | Day 1 through end of infusion with minocycline
  Concomitant antibiotics include those used between the first and last dose of minocycline IV. The number of participants and the type of antibiotic taken will be presented.
Proportion Of Participants With A Clinical Outcome Of Cure, Improved, Or Failure | Up to 30 days after minocycline infusion
  Clinical assessments will be based on participant records between end of infusion to 30 days following the last dose of minocycline (includes minocycline IV plus oral minocycline). Clinical categories for assessment include:
  * Cure: Clinical signs and symptoms are resolved and no additional antibiotic therapy is necessary for the treatment of the infection
  * Improved: Partial resolution of clinical signs and symptoms and no additional antibiotic therapy is necessary for the treatment of the infection
  * Failure: Inadequate resolution, or new or worsening clinical signs and symptoms, such that additional antibiotic therapy is necessary for treatment of the infection
  * Non-evaluable: Unable to determine response because the participant record did not contain the necessary information to determine cure, improvement, or failure.
Proportion Of Participants With A Microbiologic Eradication Or Microbiologic Persistence | Up to 30 days after minocycline infusion
  Microbiological assessments will be based on participant records between end of infusion to 30 days following the last dose of minocycline (includes minocycline IV plus oral minocycline). Microbiological categories will include only gram-negative pathogens believed to be related to the primary infection and are defined as:
  * Eradication: Documentation of a negative bacterial culture from the same site as the initial positive baseline culture
  * Presumed eradication: The absence of follow-up microbiological data/information in a participant with a clinical response of cure or improved
  * Persistence: Bacterial growth from the same site as the initial positive baseline culture excluding colonization; also referred to as microbiologic failure.

CONTACTS AND LOCATIONS:
Overall Officials: Medical Information, Study Director — Melinta Therapeutics
Locations (6):
- United States (6):
  - Lee Memorial Health System, Fort Myers, Florida
  - Florida Hospital Orlando, Orlando, Florida
  - University Medical Center of Southern Nevada, Las Vegas, Nevada
  - Maimonides Medical Center, Brooklyn, New York
  - Infectious Disease and Pulmonary Consultant, Victoria, Texas
  - University of Utah Health Sciences Center, Salt Lake City, Utah

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Minocycline Intravenous for the Treatment of Serious Infections Due to Gram-Negative Nonpseudomonal Bacteria, Including Stenotrophomonas maltophilia, Acinetobacter baumannii, and Burkholderia cepacia — https://journals.lww.com/infectdis/Fulltext/2020/07000/Minocycline_Intravenous_for_the_Treatment_of.8.aspx
- Available data/document: Package Insert: MINOCIN® (minocycline) — http://www.minociniv.com/pdfs/minocin-us-prescribing-information.pdf — MINOCIN® (minocycline) for Injection 100 mg/vial. United States Prescribing Information.